CLINICAL TRIAL: NCT00600470
Title: Collaborative Mental Health Services for Behavior Disorders in Primary Care
Brief Title: Effectiveness of Collaborative Services in Primary Care for Treating Children With Behavior Disorders
Acronym: SKIP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Kolko, Professor of Psychiatry, Psychology, and Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH063272 (NIH); R01MH063272 (NIH); DSIR 84-CTS
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders
Keywords: Behavior Problems; Behavior Disorders
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Doctor-office collaborative care management
  Interventions: Behavioral: Doctor-office collaborative care (DOCC) management
- 2 (Active Comparator): Treatment as usual: psychoeducation and outside referral to treatment (PORT). In papers, this arm is referred to as "Enhanced Usual Care (EUC)".
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Doctor-office collaborative care (DOCC) management — DOCC is an evidence-based psychosocial treatment approach that incorporates (1) adaptation of an evidence-based collaborative care approach using the chronic care model and participatory management theory to enhance training, implementation, and sustainability; (2) revised protocol content that includes medication management for ADHD, brief anxiety management, and attention to parental/partner dysfunction; (3) technological developments to facilitate screening/assessment, monitoring, and communication; and (4) an improved methodology that includes new samples, measures, and settings.
  Other Names: DOCC
  Arms: 1
Behavioral: Treatment as usual (TAU) — TAU involves routine care: psychoeducation and referral to outside providers.
  Other Names: PORT
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a doctor-office collaborative care approach in treating children with disruptive behavior problems in the pediatric primary care setting.

DETAILED DESCRIPTION:
Disruptive behavior problems (DBP) involve a behavioral tendency of children and adolescents to continually disregard basic social rules and the rights of others. Symptoms of DBP include problematic aggression, antisocial tendencies, serious defiance of rules, and temper tantrums. Children or adolescents with DBP display this type of behavior at school, home, or other social situations, often affecting family life, academic performance, and relations with others. The causes of DBP are believed to be both environmental and biological. Children most at risk for DBP are those who have low birth weight, attention deficit hyperactivity disorder (ADHD), or a history of abuse or neglect. Behavioral therapy that targets parent and child skills has shown to be the most effective treatment for DBP. This study will evaluate the effectiveness of a doctor-office collaborative care (DOCC) approach in treating children with DBP in the pediatric primary care setting. The study is a continuation and extension of the parent study, Services for Kids in Primary Care (SKIP).

Participants in this single blind study will be randomly assigned to one of two treatment groups: doctor-office collaborative care (DOCC) or treatment as usual (TAU). Treatment will take place at one of eight participating primary care practices, each randomly assigned to either DOCC or TAU. All participants will undergo an initial assessment that will include a clinical evaluation with the care manager and research questionnaires. The families participating in the practices assigned to DOCC will receive cognitive behavioral therapy (CBT), parent management training (PMT), and ADHD management training. Participants will also complete ongoing behavioral questionnaires. There will be on average 12 DOCC sessions, lasting between 30 and 90 minutes, held in the primary care office. The sessions will occur over a 3- to 6-month period. The families participating in the practices assigned to TAU will receive a full review of initial assessment findings and specific recommendations for services in the community that would meet the clinical needs of the child participant. The parent/guardian of the child will also be provided psychoeducational resources via Web sites, literature, or reference materials. Lastly, participants in TAU will receive a follow-up call between 2 and 4 weeks after the initial assessment to assist with finding community programs or additional resource identification. All participants in both groups will undergo follow-up assessments at Months 6, 12, 18, 24, and 30 after the initial assessment. Each assessment will last 2 to 3 hours and will include self-report and interview questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Score of 75% on externalizing scale of PSC-17: score less than or equal to 6
* Parent/guardian is concerned about the child's mental health
* At least one parent/guardian who resides with the child is willing to participate in services and has signed an informed consent giving permission for the child to participate

Exclusion Criteria:

* Child is currently prescribed and taking any of the following medications: SSRI, neuroleptics, antidepressants.
* Emergent psychiatric conditions that require additional treatments (e.g., eating disorder/anorexia nervosa, substance dependence, PTSD-active phase, OCD, PDD/Autism/Aspergers)
* Child has current suicidal or homicidal ideation with intent and a plan
* Participation in ongoing outpatient services and plans to continue

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 858 (Actual)
Dates: Start 2000-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Vanderbilt Parent ADHD Rating Scale; Child Health and Illness Profile; Pediatric Quality of Life Inventory; Individualized Goal Attainment Rating | Measured at baseline and at Months 6, 12, 18, 24, and 30

SECONDARY OUTCOMES:
Parenting Stress Index; Brief Symptom Inventory; Alabama Parenting Questionnaire; Services Assessment for Children and Adolescents | Measured at baseline and at Months 6, 12, 18, 24, and 30

CONTACTS AND LOCATIONS:
Overall Officials: David J. Kolko, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic (WPIC), Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kolko DJ, Campo J, Kilbourne AM, Hart J, Sakolsky D, Wisniewski S. Collaborative care outcomes for pediatric behavioral health problems: a cluster randomized trial. Pediatrics. 2014 Apr;133(4):e981-92. doi: 10.1542/peds.2013-2516. Epub 2014 Mar 24. PMID 24664093